CLINICAL TRIAL: NCT04216381
Title: Multi-Institutional Validation of Trauma Specific Frailty Index
Brief Title: Trauma Specific Frailty Index
Acronym: TSFI
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 048.TRA.2019.D
Record Dates: First submitted 2019-09-12; First posted 2020-01-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-08

CONDITIONS: Physical Trauma
Keywords: geriatric
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trauma Specific Frailty Index Questionnaire — questionnaire to assess patient's pre-injury health condition
  Other Names: Trauma Specific Frailty Index

SUMMARY:
Increasing age is a known predictor of morbidity and mortality after a traumatic injury with worst outcomes seen in patients with age greater than 65 years. Geriatric trauma patients are a unique cohort of patients who are highly prone to develop decompensated state following the stress of traumatic event leading to adverse outcomes. In a prospective study the primary site demonstrated the presence of frailty syndrome as a better predictor of in-hospital complications and adverse discharge disposition among geriatric trauma patients than age. Presently, Methodist Dallas Medical Center aims to participate in the large scale prospective multi-institutional validation of TSFI to assess the sensitivity and specificity of Trauma Specific Frailty Index in predicting adverse outcomes through a diverse account utilizing multiple facilities.

DETAILED DESCRIPTION:
In the U.S, the geriatric population is the fastest growing age group. By the end of next decade, it will comprise about 20% of the total population. Frailty is a major health burden in older people. It is defined as a condition of reduced resistance to stressors, due to a decline in physiological reserves. Multiple studies have shown that frailty is associated with adverse health outcomes, such as mortality, in-hospital complications, readmissions, and adverse discharge disposition. The concept of frailty and frailty index has been implemented widely across surgical specialties to predict post-operative outcomes and mortality in aging patients.

Increasing age is a known predictor of morbidity and mortality after a traumatic injury with worst outcomes seen in patients with age greater than 65 years. Geriatric trauma patients are a unique cohort of patients who are highly prone to develop decompensated state following the stress of traumatic event leading to adverse outcomes. In a prospective study the primary site demonstrated the presence of frailty syndrome as a better predictor of in-hospital complications and adverse discharge disposition among geriatric trauma patients than age. Most of the frailty scales that exist are extensive and time consuming and their implementation in geriatric trauma patient is not feasible. To facilitate the clinical implementation of frailty in trauma Belal et al. developed the Trauma Specific Frailty Index (TSFI), which consists of 15 variables that can reliably predict the presence of frailty and pre-frailty syndrome in geriatric trauma patients. This index was based on the Rockwood CSHA frailty, which is based on deficit accumulation. In the prospective validation study of our TSFI, the 15-variable TSFI was an independent predictor adverse discharge disposition (i.e. mortality or discharge to skilled nursing facility) in geriatric trauma patients as well as adverse complications and failure to rescue. Presently, Methodist Dallas Medical Center aims to participate in the large scale prospective multi-institutional validation of TSFI.

In this prospective observational study, MDMC will participate as a site contributing to the multi-center study under the direction of Dr. Bellal at the University of Arizona. At our site, Dr. Amos will serve as site-PI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Diagnosis of physical trauma

Exclusion Criteria:

* Refusal of consent.
* Non-responsive patients who are unable to consent with no relative/proxy available to consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients ≥65 years of age who admitted with a diagnosis of physical trauma between August 2019 through August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Mortality | August 2019 through August 2020
  death of the participant
complications | August 2019 through August 2020
  complications associated with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Amos, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided